CLINICAL TRIAL: NCT01115374
Title: Efficacy of Low Frequency Sound Waves in the Treatment of Breast Cancer Related Lymphedema: a Cross-over Randomized Trial
Brief Title: Lymphedema Therapy With Sound Wave Lymphatic Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion IMIM (Other)
Responsible Party: Principal Investigator, Roser Belmonte, MD, Fundacion IMIM
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LES_OBSF_DLM
Record Dates: First submitted 2010-03-30; First posted 2010-05-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- manual lymphatic drainage (Active Comparator): Application of manual lymphatic drainage
  Interventions: Procedure: Manual lymphatic drainage
- low frequency sound waves (Experimental): Application of low frequency sound waves
  Interventions: Device: low frequency sound waves

INTERVENTIONS:
Procedure: Manual lymphatic drainage — Application of manual lymphatic drainage (one session every work day during two weeks, total 10 sessions)
  Other Names: Decongestive physiotherapy
  Arms: manual lymphatic drainage
Device: low frequency sound waves — Application of low frequency sound waves (one session every work day during two weeks, total 10 sessions)
  Other Names: Device based physiotherapy
  Arms: low frequency sound waves

SUMMARY:
Lymphedema is a frequent sequela of breast cancer treatment, that can develop up to 40% of patients. Lymphedema is the accumulation of protein-rich fluid (lymph) in the interstitial spaces of the affected body part due to a blockage or malfunction in the lymph system. It can appear in the arm, shoulder, breast, or thoracic area. Lymphedema swelling causes discomfort and sometimes disability. The treatment of lymphedema associated with breast cancer can include complex decongestive physiotherapy, compression therapy, therapeutic exercises, and pharmacotherapy.

In this study two treatments will be compared to reduce lymphedema: the manual lymphatic drainage (standard care) versus the low frequency sound waves.

DETAILED DESCRIPTION:
Lymphedema, a sequela of breast cancer and breast cancer therapy, changes functional abilities and may affect a patient's psychosocial adjustment and overall quality of life. Lymphedema is the accumulation of lymph fluid in the interstitial space. Fluid accumulation in the limbs causes enlargement, often with a feeling of heaviness.Chronic inflammation leads to fibrosis of the lymphatics, which compounds the problem. Several studies have examined the incidence of lymphedema when axillary radiation is given after axillary dissection vs radiation to an undissected axilla. The risk of lymphedema is higher in women treated with axillary dissection and adjuvant radiation to the axilla, with edema reported in 9% to 40% of patients. Patients with lymphedema may report symptoms such as a sensation of arm fullness and mild discomfort, which are seen in the early stages of the condition. Joint immobility, pain, and skin changes are noted frequently in the later stages of lymphedema. Patients also may be predisposed to infections involving the affected extremity. The treatment of lymphedema associated with breast cancer can include complex decongestive physiotherapy, compression therapy, therapeutic exercises, and pharmacotherapy. Manual lymphatic drainage is the standard decongestive therapy. Recently, low frequency sound waves has been used to reduce lymphedema. The aim of this study is to compare the efficacy of the manual lymphatic drainage versus the low frequency sound waves.

ELIGIBILITY:
Inclusion Criteria:

* Lymphedema presence at least for 1 year
* No previous treatments for lymphedema in the last 6 months

Exclusion Criteria:

* Electronic devices or metalic implants
* Cardiac failure or hypertension
* Epilepsy
* Local infection
* Pregnancy
* Thrombophlebitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Volume of lymphedema | 2 months
  Evaluation of the lymphedema volume measuring size of the extremity affected

SECONDARY OUTCOMES:
Pain | 2 months
  Visual Analog Scales of pain
Quality of life | 2 months
  Quality of life using the Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer (FACT-B+4)

CONTACTS AND LOCATIONS:
Overall Officials: Roser Belmonte, MD, Principal Investigator — Hospital de la Esperanza, Barcelona, Spain
Locations (1):
- Hospital de la Esperanza, Barcelona, Spain